CLINICAL TRIAL: NCT07119229
Title: A Multicenter, Prospective Trial Evaluating the Safety and Efficacy of the Implantable Artificial Bronchus (IAB) in Adults Suffering From Severe Emphysema
Brief Title: A Multi Center Study Testing a New Implant for Adults With Severe Emphysema
Acronym: IAB-2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pulmair Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAB2-CIP-v01
Record Dates: First submitted 2025-07-28; First posted 2025-08-13 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Emphysema or COPD; Emphysema; COPD
Keywords: IAB; Stent; Emphysema treatment; emphysema study; COPD treatment; COPD study; EBV alternative; Lung volume reduction; Lung hyperinflation treatment
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- All subjects will receive study treatment (Experimental): All subjects will receive treatment with a maximum of 10 Implantable Artificial Bronchus (IABs) which are polymer based stents that can be permanently placed in any diseased lobe of the lungs.
  Interventions: Device: Implantable Artificial Bronchus

INTERVENTIONS:
Device: Implantable Artificial Bronchus — The Implantable Artificial Bronchus (IAB) is a tapered, flexible and fenestrated polymer-based airway stent that is implanted bronchoscopically using a proprietary delivery system into diseased lungs of patients with emphysema.
  Other Names: IAB

SUMMARY:
A study taking place at multiple sites in the United States, Europe and Brazil to evaluate how well a new therapy for severe COPD/emphysema works, and how safe it is.

DETAILED DESCRIPTION:
IAB-2 is an open-label (unblinded), multicenter, prospective trial of the Implantable Artificial Bronchus (IAB) in adults suffering from severe COPD/emphysema. There is no control group or comparator. The study will be conducted at as many as twelve sites in the United States and three sites outside of the US, in the Netherlands, Germany and Brazil.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent.
2. Diagnosis of COPD/emphysema.
3. At least 22-years of age.
4. 18 ≤ BMI ≤ 32.
5. 6-minute walk Distance between 100-meters and 400-meters at baseline exam.
6. Stable disease with less than 10-mg prednisone (or equivalent) daily
7. Non-smoking for 4-months prior to screening interview (including tobacco, vaping, marijuana, etc.).
8. FEV1 between 15% and 50% of predicted value at baseline exam.
9. FEV1/FVC <70%.
10. Subject has ≥25% emphysema destruction score in each lung defined by areas of low attenuation <-950 HU, as determined by CT core lab.
11. Subject has homogeneous or heterogeneous emphysema, and at least one lung has a 15% difference between upper and lower lobes in emphysema destruction score (< -950HU) as determined by CT core lab.
12. RV > 175% of predicted value.
13. mMRC score ≥ 2.

Exclusion Criteria:

* 1. Currently participating in another clinical study that involves surgery, interventional or pharmaceutical treatment..

  2. α-1 Antitrypsin deficiency 3. Women of child-bearing potential. 4. More than 2 COPD exacerbation episodes requiring hospitalization in the last year prior to screening.

  5. Any COPD exacerbations requiring hospitalization within 6-weeks of planned intervention.

  6. Two or more instances of pneumonia episodes requiring hospitalization in the last year prior to screening.

  7. Clinically significant mucus production or chronic bronchitis. 8. Myocardial Infarction or unstable / uncontrolled congestive heart failure within 6-months of screening.

  9. Prior lung transplant, LVRS, bullectomy, lobectomy or endoscopic lung volume reduction (ELVR).

  10. Clinically significant bronchiectasis. 11. Unable to safely discontinue anti-coagulants or platelet activity inhibitors for 7-days.

  12. Uncontrolled pulmonary hypertension (systolic pulmonary arterial pressure >45 mm Hg) or evidence or history of cor pulmonale as determined by recent echocardiogram (completed within the last 3-months prior to screening visit). Note: the echocardiogram is not a required screening procedure.

  13. Suspected malignant pulmonary nodule or other lung cancer. 14. HRCT collected per CT scanning protocol within the last 6-months of screening date and evaluated by clinical site personnel using 3D segmentation software shows:
  1. Large bullae encompassing greater than 30% of either lung
  2. Insufficient landmarks to evaluate the CT study using the software as it is intended
  3. All lobes are less than 25% parenchyma diseased (< -950 HU) 15. Any cardiac comorbidity which the PI believes would compromise the safety of the patient after an IAB implant.

     16. TLC < 100% predicted at screening. 17. DLCO < 15% or > 50% of predicted value at screening. 18. PaCO2 > 50 mm Hg at screening. 19. PaO2 < 45 mm Hg in room air at screening. 20. Plasma cotinine level > 13.7 ng/ml or carboxyhemoglobin (arterial or ear lobe capillary) >2.5% at screening.

     21. Current diagnosis of substance abuse disorder. 22. Current diagnosis of any of the following: Major Depressive Disorder (MDD), Schizoaffective Disorder, Schizophrenia, Borderline Personality Disorder, Bipolar Disorder.

     23. Any other conditions, which, in the opinion of the Investigator, would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Absolute change in residual volume (RV) | 90 days after last IAB is implanted
  The primary endpoint is the absolute change in residual volume (RV) from baseline to endpoint as recorded 90-days after the last implant.

SECONDARY OUTCOMES:
Changes from baseline to 90-days, involving pulmonary function, exercise tolerance, dyspnea burden and occurrence as well as all related adverse device effects | 90 days after last implant
  Absolute change in Forced Expiratory Volume in one second (FEV1) from baseline to endpoint; Absolute change in residual volume/total lung capacity (RV/TLC) from baseline to endpoint; Absolute change in Six-minute Walk Distance (6MWD); Absolute change in the St George's Respiratory Questionnaire (SGRQ) total score where a higher score represents more significant impact of the disease on wellbeing; Absolute change in the Modified Medical Research Counsel Questionnaire (mMRC) dyspnea score; Absolute changes in COPD Assessment Test (CAT), with higher scores indicating a greater impact of COPD on health; Absolute change in EQ-5D Summary Index Questionnaire which measures self-reported assessment of mobility, self-care, usual activities, pain/discomfort and anxiety/depression with a higher score indicating more significant impact of the disease on each dimension.
  Adverse Device Effects (ADEs), Serious Adverse Device Effects (SADEs) and Device Deficiencies (DDs) with SADE potential

CONTACTS AND LOCATIONS:
Overall Officials: George Cheng, MD, PhD., Principal Investigator — Unversity of California San Diego

IPD SHARING:
Plan to Share IPD: No